CLINICAL TRIAL: NCT03073525
Title: A Randomized, Intra-patient Crossover, Safety, Biomarker and Anti-Tumor Activity Assessment of the Combination of Atezolizumab and Vigil in Patients With Advanced Gynecological Cancers (A Companion Study to CL-PTL-119)
Brief Title: A Trial of Atezolizumab and Vigil in Patients With Advanced Gynecological Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-126
Expanded Access: NCT03842865 (Temporarily not available)
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Advanced Gynecological Cancers; Ovarian Cancer; Cervical Cancer; Uterine Cancer
Keywords: Stage IIIb; Stage IV; Ovarian Cancer; Cervical Cancer; Uterine Cancer; Immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — FANG vaccine; atezolizumab

STUDY DESIGN:
Intervention Model Description: This was a 3 part study. Parts 1 and 3 did not involve randomization. In part 2, eligible participants were randomized to receive two cycles of either Vigil alone or Atezolizumab alone, then followed by combination treatment with the two agents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Vigil + Atezo (Experimental): This was a safety run in and intervention was combined. The first three participants received Vigil immunotherapy at a concentration of 1x10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks. 1 cycle = 21 days.
  Interventions: Biological: Vigil; Drug: Atezolizumab
- Part 2: Vigil first then combination Vigil + Atezo (Experimental): After Part 1 participants completed completed combination therapy without dose-limiting toxicity, then Part 2 participants randomized to Vigil first received two cycles of Vigil alone, then Vigil and atezolizumab given in sequence (Vigil administered first, followed 30 minutes later by atezolizumab)
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 107 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil
  1 cycle = 21 days
  Interventions: Biological: Vigil; Drug: Atezolizumab
- Part 2: Atezo first then combination of Vigil + Atezo (Experimental): After Part 1 participants completed completed combination therapy without dose-limiting toxicity, then Part 2 participants randomized to atezolizumab first received two cycles of atezolizumab alone, then Vigil and atezolizumab given in sequence (Vigil administered first, followed 30 minutes later by atezolizumab).
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 107 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. 1 cycle = 21 days
  Interventions: Biological: Vigil; Drug: Atezolizumab
- Part 3: Atezo Only (Other): Participants who completed all cycles of Part 2 were pre-approved by the sponsor for inclusion into Part 3. Atezolizumab alone was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks. 1 cycle = 21 days
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Biological: Vigil — The Vigil vaccine is made up of irradiated autologous tumor cells which have been electroporated ex vivo with the Vigil plasmid designed to suppress expression of both the TGFβ1 and TGFβ2 proteins while simultaneously expressing rhGMCSF protein.
  Other Names: Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy; FANG vaccine
  Arms: Part 1: Vigil + Atezo; Part 2: Atezo first then combination of Vigil + Atezo; Part 2: Vigil first then combination Vigil + Atezo
Drug: Atezolizumab — Atezolizumab was prepared and administered at the FDA approved dose and schedule as described in the U.S. Package Insert (USPI). The initial dose was administered over one hour and if well tolerated, subsequent infusions may have been administered over 30 minutes.
  Atezolizumab in formulation F03 (1200 mg per vial) was administered in 250 mL 0.9% NaCl IV infusion bags and infusion lines equipped with 0.2 μm in-line filters.
  Other Names: TECENTRIQ™; MPDL3280A

SUMMARY:
The clinical trial was a companion study to protocol CL-PTL-119 (A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial of Vigil Engineered Autologous Tumor Cell Immunotherapy in Subjects with Stage IIIb-IV Ovarian Cancer in Clinical Complete Response following Surgery and Primary Chemotherapy (VITAL) NCT02346747). Participants who had investigational product (Vigil) successfully made but were not eligible to enroll onto the VITAL study or previously randomized to placebo were given the opportunity to participate in this protocol. The main goal of this clinical trial was to determine the safety of combining Vigil therapy with atezolizumab.

DETAILED DESCRIPTION:
The clinical trial was intended as a companion study to protocol CL-PTL-119 (VITAL study; NCT 02346747). Subjects who had tumor harvested at surgery and Vigil successfully manufactured, but then were ineligible for randomization onto the VITAL study or previously randomized to placebo, and also in subjects who have recurrent ovarian cancer were offered the opportunity to participate in this protocol. The trial was a multi-center, randomized, 3-part, open label study of Vigil, the checkpoint inhibitor atezolizumab and the combination of the two agents, in subjects with treatment refractory or recurrent epithelial ovarian cancer, or other gynecological cancers (i.e., cervical, uterine).

Part 1 was a safety run-in cohort and intervention (Vigil plus atezolizumab) was combined. The first 3 subjects registered in the trial were assigned to Part 1.

Part 2 was conducted after Part 1 participants completed combination therapy without dose-limiting toxicity. The purpose of Part 2 was to determine if Vigil given first then in sequence with atezolizumab would enhance immunotherapeutic anticancer activity. The overall efficacy of administration sequence was assessed.

Eligible subjects were randomized to receive two cycles of Vigil alone (n= 11) or two cycles of atezolizumab alone (n=10), followed by combination treatment with both of the agents.

Part 3 was an expansion cohort to allow subjects who completed all cycles of Part 2 to continue on atezolizumab alone, after Cycle 12. In this study, only 1 subject from Part 2 received additional treatment with atezolizumab. Pre-approval by sponsor was required by the sponsor before allowing subjects to continue treatment with atezolizumab in Part 3.

Subjects remained on treatment until disease progression or death or product toxic effect. Disease progression was determined radiographically by local investigators using the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

Part 1, radiological assessment of tumor response was performed at baseline and every third cycle thereafter. Tumor biopsy for correlative studies including scoring of tumor infiltrating lymphocyte (TIL) and PD-1 / PD-L1 expression analysis was obtained at tissue procurement and at any time after the end of cycle 3. Whole blood for correlative studies (immune function) was obtained at baseline, prior to study agent administration at the start of cycle 3 and every third cycle thereafter.

Part 2, radiological assessment of tumor response was performed at baseline, at the end of cycle 2 of single agent therapy, and every third cycle thereafter. Tumor biopsy for correlative studies including scoring of tumor infiltrating lymphocyte (TIL) and PD-1 / PD-L1 expression analysis was obtained at tissue procurement, prior to the start of combination therapy and at any time after the end of cycle 3. Whole blood for correlative studies (immune function) was obtained at baseline, prior to study agent administration at the start of cycle 3 (the first cycle of combination therapy) and every third cycle thereafter.

Part 3 schedule of assessments continued from Part 2 in which the following was assessed every third cycle: radiological assessments, tumor biopsy (if available), and whole blood collection for correlative studies.

The safety evaluation included recording of AEs and SAEs, and changes from baseline in laboratory evaluations, vital signs, electrocardiograms, and physical examinations.

Treatment was administered on an outpatient basis. A study cycle is defined as 21 days (3 weeks). Treatment was allowed to continue unless documented disease progression, discontinuation for toxicity, withdrawal of consent, or meeting other criteria for withdrawal from study. After progression, participants were contacted annually for three years for documentation of survival status information.

ELIGIBILITY:
Tissue Procurement Inclusion Criteria:

Subjects will be eligible for tissue procurement for the Vigil manufacturing process, if they meet all of the following criteria:

1. Histologically confirmed Stage IIIb, IIIc or IV high-grade papillary serous, clear cell, or endometrioid ovarian, fallopian tube or primary peritoneal carcinoma
2. Age ≥ 18 years.
3. Estimated survival ≥ 6 months.
4. ECOG Performance Status ≤ 1
5. Metastatic disease
6. Planned standard of care surgical procedure (e.g., tumor biopsy or palliative resection or thoracentesis) and expected availability of a cumulative soft-tissue mass of ~10-30 grams tissue ("grape" to "golf-ball" size) or ascites fluid estimated volume ≥ 500mL (from a primary or secondary paracentesis, yielding in a high volume of tumor cells) for immunotherapy manufacture.
7. Tumor intended for immunotherapy manufacture is not embedded in bone and does not contain luminal tissue (e.g. bowel, ureter, bile duct).
8. Ability to understand and the willingness to sign a written informed protocol specific consent for tissue harvest or a parental/guardian informed consent and pediatric assent when appropriate.

Tissue Procurement Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for tissue procurement for the Vigil manufacturing:

1. Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily) for < 30 days duration.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
3. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
4. Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids.
5. Known HIV or chronic Hepatitis B or C infection.
6. Known history of allergies or sensitivities to gentamicin.
7. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
8. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) less than 21 days prior to tissue procurement.

Study Enrollment Inclusion Criteria:

Subjects will be eligible for registration into the trial if they meet all of the following inclusion criteria:

1. Successful manufacturing of at least 4 vials of Vigil.
2. One of the following:

   1. Failure to meet the eligibililty criteria for Protocol CL-PTL-119 due to i) histology of ovarian cancer and failure to achieve a complete clinical response following primary debulking surgery and standard paclitaxel/carboplatin therapy OR, ii) a histologic diagnosis of another gynecologic malignancy which is not ovarian cancer.
   2. Recurrent ovarian cancer.
   3. Randomized on Protocol CL-PTL-119 and were subsequently unblinded at recurrence and were assigned to the placebo arm.
3. ECOG performance status (PS) ≤ 1 (or ≤ 2 due to carcinoid syndrome).
4. Estimated survival ≥ 6 months.
5. Measureable per RECIST 1.1 or evaluable disease.
6. Adequate organ and bone marrow function as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10e9/L (1500 per mm^3)
   2. Platelets >100 × 10e9/L (100,000 per mm^3)
   3. Hemoglobin ≥9.0 g/dL (5.59 mmol/L)
   4. Creatinine clearance (CrCL) >50 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance:

      Females:

      CrCL (mL/min) = Weight (kg) × (140 - Age) × 0.85/72 × serum creatinine (mg/dL)
   5. Serum bilirubin ≤1.5 × upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of hemolysis or hepatic pathology) who will be allowed in consultation with their physician.
   6. AST and ALT ≤2.5 × ULN in patients with no liver metastasis
   7. AST or ALT ≤5 × ULN in patients with liver metastasis
   8. TSH within institutional limits. If TSH is greater or less than institutional limits patients may participate if their T4 is within normal limits (WNL); patients may be on a stable dose of replacement thyroid medication; dose adjustments are allowed if needed
7. Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery (or ≤ 2 due to carcinoid syndrome).
8. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade 2 or better
9. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the IPs (Vigil and/or atezolizumab) may be included (e.g., hearing loss) after consultation with the Principal Investigator
10. Subjects who are not rendered surgically sterile as a result of surgery for ovarian cancer, must have, negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
11. Ability to understand and the willingness to sign a written informed protocol specific consent.
12. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up. Patients must have fully recovered from chemotherapy associated toxicities prior to starting treatment on this protocol.
13. Palliative radiotherapy is permitted provided:

    1. More than 3 weeks have elapsed between the end of radiotherapy and the first dose of study therapy, AND
    2. The irradiated lesion(s) (unless measurable progression after irradiation) cannot be used as target lesions.

Study Enrollment Exclusion Criteria:

In addition to the procurement exclusion, subjects (both with Vigil manufactured and undergoing procurement) will NOT be eligible for study registration and enrollment if meeting any of the following criteria:

1. Participation in another clinical study with an investigational product within the last 3 weeks prior to study start.
2. Receipt of steroid therapy within the 2 weeks of the first dose of study therapy.
3. Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy. NOTE: Subjects, if enrolled, should not receive live vaccine during the study and for 5 months after the last dose of atezolizumab.
4. Post-surgery complication that in the opinion of the treating investigator would interfere with the subject's study participation or make it not in the best interest of the subject to participate.
5. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
6. Female subjects who are pregnant, breast-feeding or of reproductive potential who are not employing an effective method of birth control defined in the protocol. Effective contraception is required for women receiving atezolizumab for 5 months after the last dose.
7. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
8. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) less than 21 days prior to the first dose of study drug or less than 6 weeks for nitrosourea or mitomycin C.
9. Receipt of any anti-cancer therapy between tissue procurement on CL-PTL-126 and first dose of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (6):
- United States (6):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Billings Clinic, Billings, Montana
  - Dartmouth-Hitchcock Medical Center/ Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Prisma Health Cancer Institute, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Senzer N, Barve M, Nemunaitis J, Kuhn J, Melnyk A, et al. (2013) Long Term Follow Up: Phase I Trial of "Bi-Shrnafurin/GMCSF DNA/Autologous Tumor Cell" Immunotherapy (FANG™) in Advanced Cancer. J Vaccines Vaccin 4:209. doi:10.4172/2157-7560.1000209
- [Background] Rocconi RP, Grosen EA, Ghamande SA, Chan JK, Barve MA, Oh J, Tewari D, Morris PC, Stevens EE, Bottsford-Miller JN, Tang M, Aaron P, Stanbery L, Horvath S, Wallraven G, Bognar E, Manning L, Nemunaitis J, Shanahan D, Slomovitz BM, Herzog TJ, Monk BJ, Coleman RL. Gemogenovatucel-T (Vigil) immunotherapy as maintenance in frontline stage III/IV ovarian cancer (VITAL): a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Oncol. 2020 Dec;21(12):1661-1672. doi: 10.1016/S1470-2045(20)30533-7. PMID 33271095
- [Background] Oh J, Barve M, Senzer N, Aaron P, Manning L, Wallraven G, Bognar E, Stanbery L, Horvath S, Manley M, Nemunaitis J, Walter A, Rocconi RP. Long-term follow-up of Phase 2A trial results involving advanced ovarian cancer patients treated with Vigil(R) in frontline maintenance. Gynecol Oncol Rep. 2020 Sep 17;34:100648. doi: 10.1016/j.gore.2020.100648. eCollection 2020 Nov. No abstract available. PMID 33364285
- [Background] Rocconi RP, Monk BJ, Walter A, Herzog TJ, Galanis E, Manning L, Bognar E, Wallraven G, Stanbery L, Aaron P, Senzer N, Coleman RL, Nemunaitis J. Gemogenovatucel-T (Vigil) immunotherapy demonstrates clinical benefit in homologous recombination proficient (HRP) ovarian cancer. Gynecol Oncol. 2021 Jun;161(3):676-680. doi: 10.1016/j.ygyno.2021.03.009. Epub 2021 Mar 11. PMID 33715892
- [Result] Rodney Paul Rocconi, Erin E. Stevens, Justin N. Bottsford-Miller, Sharad A. Ghamande, Phylicia Aaron, Gladice Wallraven, Ernest Bognar, Meghan Manley, Staci Horvath, Luisa Manning, John J. Nemunaitis, Thomas J Herzog, Bradley J. Monk, Robert L. Coleman, and Vigil Team (2020), A phase I combination study of vigil and atezolizumab in recurrent/refractory advanced-stage ovarian cancer: Efficacy assessment in BRCA1/2-wt patients. DOI: 10.1200/JCO.2020.38.15_suppl.3002 Journal of Clinical Oncology 38, no. 15_suppl (May 20, 2020) 3002-3002.
- [Result] Rocconi RP, Stevens EE, Bottsford-Miller JN, Ghamande SA, Elder J, DeMars LL, Munkarah A, Aaron P, Stanbery L, Wallraven G, Bognar E, Manley M, Horvath S, Manning L, Walter A, Galanis E, Herzog T, Monk BJ, Coleman RL, Nemunaitis J. Proof of principle study of sequential combination atezolizumab and Vigil in relapsed ovarian cancer. Cancer Gene Ther. 2022 Mar;29(3-4):369-382. doi: 10.1038/s41417-021-00317-5. Epub 2021 Mar 22. PMID 33753870

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-five (25) subjects signed the informed consent to enter the treatment portion of the trial. One (1) subject was ineligible, and a total of 24 subjects received treatment in the study.
Groups:
- Part 1: Vigil + Atezo: This was a safety run in and intervention was combined. The first three participants received Vigil immunotherapy at a concentration of 1x10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks. Vigil was administered first, followed 30 minutes later by atezolizumab. 1 cycle = 21 days.
- Part 2: Vigil Then Vigil + Atezo: After Part 1 participants completed combination therapy without dose-limiting toxicity, then Part 2 participants randomized to Vigil first received two cycles of Vigil alone, then Vigil and atezolizumab given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab.
  Participants who completed all cycles of Part 2 were pre-approved by the sponsor for inclusion into Part 3. Atezolizumab alone was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks.
  1 cycle = 21 days
- Part 2: Atezo Then Vigil + Atezo: After Part 1 participants completed combination therapy without dose-limiting toxicity, then Part 2 participants randomized to atezolizumab first received two cycles of atezolizumab alone, then Vigil and atezolizumab given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab.
  Participants who completed all cycles of Part 2 were pre-approved by the sponsor for inclusion into Part 3. Atezolizumab alone was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks.
  1 cycle = 21 days
Period: Overall Study
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo
Started | 3 | 11 | 10
Part 3: Atezolizumab Alone (Part 3 did not apply to Participants who completed Part 1.) | 0 | 1 | 0
Completed | 3 | 11 | 7
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Number of subjects randomized with recurrent ovarian cancer or failed to meet eligibility criteria of CL-PTL-119. There was no separate analysis for Part 3 as the one subject's data was included in Part 2 analysis.
Groups:
- Part 2: Vigil Then Vigil + Atezo: After Part 1 participants completed combination therapy without dose-limiting toxicity, then Part 2 participants randomized to Vigil first received two cycles of Vigil alone, then Vigil and atezolizumab given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab.
  1 cycle = 21 days
- Part 2: Atezo Then Vigil + Atezo: After Part 1 participants completed combination therapy without dose-limiting toxicity, then Part 2 participants randomized to atezolizumab first received two cycles of atezolizumab alone, then Vigil and atezolizumab given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab. 1 cycle = 21 days
- Total: Total of all reporting groups
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo | Total
Number analyzed (Participants) | 3 | 11 | 10 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7 | 14
  >=65 years | 1 | 6 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 10 | 24
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 3 | 9 | 8 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 11 | 10 | 24
Number of Prior Lines of Systemic Therapies [Count of Participants; unit: Participants] — The number of prior lines of systemic therapies was obtained from medical records during the pre-study period. Systemic therapies refers to any type of cancer treatment that targets the entire body.
  Participants
    1 | 0 | 5 | 2 | 7
    2 | 1 | 4 | 3 | 8
    3 | 1 | 2 | 4 | 7
    4 | 1 | 0 | 1 | 2
Baseline ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Scale is a standard way of to assess how a patient with cancer is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. ECOG scores range from 0 to 5. A lower score means the patient is better able to carry out daily activities. The assessment is made during the clinical study visit.
  Participants
    0 | 2 | 7 | 2 | 11
    1 | 1 | 4 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent AEs of Vigil + Atezolizumab
Description: The safety evaluation included Adverse Events (AEs), Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs) and changes from baseline in laboratory evaluations, vital signs, electrocardiograms and physical examinations. AEs were graded according to the National Cancer Institute (NCI) CTCAE v4.03 and coded using the Medical Dictionary for Regulatory Activities. Laboratory abnormalities were graded according to the NCI CTCAE v4.03, if applicable.
Time Frame: AEs reported from first treatment dose and up to 30 days after last treatment, about 12 months.
Population: Grade 3/4 treatment-related events from first dose up to 30 days after last treatment.
Measure: Number; unit: adverse events
Groups:
- Part 2: Vigil Then Vigil + Atezo: Patients in Part 1 completed combination therapy without dose-limiting toxicity justifying expansion to Part 2. This arm was to determine if Vigil given first then combined with atezolizumab would enhance immunotherapeutic anticancer activity. Overall, efficacy of administration sequence was assessed.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab.
  1 cycle = 21 days
- Part 2: Atezo Then Vigil + Atezo: Patients in Part 1 completed combination therapy without dose-limiting toxicity justifying expansion to Part 2. This arm was to determine if atezolizumab given first then combined with Vigil would enhance immunotherapeutic anticancer activity. Overall, efficacy of administration sequence was assessed.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab. 1 cycle = 21 days
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo
Number analyzed (Participants) | 3 | 11 | 10
adverse events
  Grade 4 Atezolizumab-Related | 0 | 0 | 0
  Grade 4 Vigil-Related | 0 | 0 | 0
  Grade 3 Atezolizumab-Related | 0 | 1 | 4
  Grade 3 Vigil-Related | 0 | 0 | 0

2. Secondary Outcome: Immune Response Rate
Description: Whole blood for correlative studies will be obtained at baseline, at the start of cycle 3 (the first cycle of combination therapy), every 3 cycles thereafter and end of treatment.
Time Frame: Up to 30 days after last treatment
Population: Samples were not analyzed for immune response data.
Groups:
- Part 2: Vigil Then Vigil + Atezo: After Part 1 participants completed combination therapy without dose-limiting toxicity, Part 2 participants randomized to Vigil first received two cycles of Vigil alone, then Vigil and atezolizumab given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab.
  1 cycle = 21 days
- Part 2: Atezo Then Vigil + Atezo: After Part 1 participants completed combination therapy without dose-limiting toxicity, Part 2 participants randomized to atezolizumab first received two cycles of atezolizumab alone, then Vigil and atezolizumab given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. When Vigil and atezolizumab was given together, Vigil was administered first, followed 30 minutes later by atezolizumab. 1 cycle = 21 days
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Time to Progression
Description: Overall assessment of time to progression and survival will be measured by Radiological Tumor Assessment by local investigators using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
  In Part 1, disease progression was assessed at baseline and every third cycle thereafter. In Part 2, the disease was assessed at baseline, at the end of Cycle 2 of single-agent therapy, and every third cycle thereafter.
Time Frame: From baseline (prior to treatment) up to 3 years
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 1: Vigil + Atezo: Part 1 is a safety run-in cohort. Vigil immunotherapy will be administered at a concentration of 1x10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab will be administered at a dose of 1200 mg as an intravenous infusion every 3 weeks. The initial dose is to be administered over one hour and if well tolerated, subsequent infusions may be administered over 30 minutes. Vigil should be administered first, followed 30 minutes later by atezolizumab.
  Vigil: Vigil is composed of autologous tumor cells harvested from the patient at the time of initial de-bulking surgery which are then transfected extracorporeally, with a plasmid encoding for the gene for GM-CSF, an immune-stimulatory cytokine, and a bifunctional, short hairpin RNA which specifically knocks down the expression of furin, the critical convertase responsible for production of the two TGβ isoforms (TGFβ-1 and TGFβ-2).
  Atezolizumab: Atezolizumab is provided in a single-use, 20-cc USP/Ph. Eur. Type 1 glass vial as a colorless to slightly-yellow, sterile, preservative-free clear liquid solution intended for IV administration. The vial is designed to deliver 20 mL (1200 mg) of atezolizumab solution but may contain more than the stated volume to enable delivery of the entire 20 mL volume. The atezolizumab drug product is formulated as 60 mg/mL atezolizumab in 20 mM histidine acetate, 120 mM sucrose, 0.04% polysorbate 20, pH 5.8.
- Part 2: Vigil Then Vigil + Atezo: Part 2 is a randomized, open label study of Vigil, the checkpoint inhibitor Atezolizumab and the combination of the two agents.
  Vigil immunotherapy will be administered at a concentration of 1x10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses for 2 cycles (1 cycle = 21 days).
  Vigil: Vigil is composed of autologous tumor cells harvested from the patient at the time of initial de-bulking surgery which are then transfected extracorporeally, with a plasmid encoding for the gene for GM-CSF, an immune-stimulatory cytokine, and a bifunctional, short hairpin RNA which specifically knocks down the expression of furin, the critical convertase responsible for production of the two TGβ isoforms (TGFβ-1 and TGFβ-2).
  Atezolizumab: Atezolizumab is provided in a single-use, 20-cc USP/Ph. Eur. Type 1 glass vial as a colorless to slightly-yellow, sterile, preservative-free clear liquid solution intended for IV administration. The vial is designed to deliver 20 mL (1200 mg) of atezolizumab solution but may contain more than the stated volume to enable delivery of the entire 20 mL volume. The atezolizumab drug product is formulated as 60 mg/mL atezolizumab in 20 mM histidine acetate, 120 mM sucrose, 0.04% polysorbate 20, pH 5.8 (Phase III formulation).
- Part 2: Atezo Then Vigil + Atezo: Part 2 is a randomized, open label study of Vigil, the checkpoint inhibitor Atezolizumab and the combination of the two agents
  Atezolizumab will be administered at a dose of 1200 mg as an intravenous infusion every 3 weeks for 2 cycles (1 cycle = 21 days). The initial dose is to be administered over one hour and if well tolerated, subsequent infusions may be administered over 30 minutes.
  Vigil: Vigil is composed of autologous tumor cells harvested from the patient at the time of initial de-bulking surgery which are then transfected extracorporeally, with a plasmid encoding for the gene for GM-CSF, an immune-stimulatory cytokine, and a bifunctional, short hairpin RNA which specifically knocks down the expression of furin, the critical convertase responsible for production of the two TGβ isoforms (TGFβ-1 and TGFβ-2).
  Atezolizumab: Atezolizumab is provided in a single-use, 20-cc USP/Ph. Eur. Type 1 glass vial as a colorless to slightly-yellow, sterile, preservative-free clear liquid solution intended for IV administration. The vial is designed to deliver 20 mL (1200 mg) of atezolizumab solution but may contain more than the stated volume to enable delivery of the entire 20 mL volume. The atezolizumab drug product is formulated as 60 mg/mL atezolizumab in 20 mM histidine acetate, 120 mM sucrose, 0.04% polysorbate 20, pH 5.8 (Phase III formulation).
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo
Number analyzed (Participants) | 3 | 11 | 10
months | 3.42 [1.61 to NA] — Not Reached | 3.42 [3.3 to NA] — Not Reached | 2.86 [2.50 to NA] — Not Reached

4. Secondary Outcome: Radiographic Overall Response Rate (ORR)
Description: Radiographic ORR is defined as the percentage of participants achieving a Complete Response (CR) or Partial Response (PR), as assessed by investigators using RECIST 1.1.
  In Part 1, ORR was assessed at baseline and every third cycle thereafter. In Part 2, the disease was assessed at baseline, at the end of Cycle 2 of single-agent therapy, and every third cycle thereafter.
  95% confidence interval from exact binomial distribution (Blopper-Pearson method).
Time Frame: From first dose to end of study treatment (up to 9 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo
Number analyzed (Participants) | 3 | 11 | 10
percentage of participants with response | 33 [0.8 to 90.6] | 9 [0.2 to 41.3] | 10 [.03 to 44.5]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time of randomization to date of death due to any cause.
Time Frame: OS will be evaluated from time of randomization up to 37 months following documented disease progression.
Population: All treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil Then Vigil + Atezo | Part 2: Atezo Then Vigil + Atezo
Number analyzed (Participants) | 3 | 11 | 10
Months | 8.2 [5.78 to NA] — Not enough patients have had an event | 37.0 [18.50 to NA] — Not enough patients have had an event | 15.1 [5.22 to NA] — Not enough patients have had an event

ADVERSE EVENTS:
Time Frame: SAEs and Other Adverse Events: Adverse events were recorded from time of first dose of Vigil and/or atezolizumab up to 30 days following the last dose of study treatment or until another therapy was initiated (up to 12 months). All-cause Mortality: from randomization and up to 37 months following disease progression.
Description: All treated participants.
Groups:
- Part 2: Vigil: Part 2 participants randomized to Vigil first received Vigil immunotherapy at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection for the first two cycles.
  1 cycle = 21 days
- Part 2: Atezo: Part 2 participants randomized to atezolizumab first received atezolizumab at a dose of 1200 mg as an intravenous infusion for the first two cycles. 1 cycle = 21 days
- Part 2: Vigil and Atezo: After Part 2 participants completed the first two cycles of Vigil or atezolizumab, then Vigil and atezolizumab was given in sequence.
  Vigil immunotherapy was administered at a concentration of 1 x 10e6 or 1 x 10e7 cells/dose given via intradermal injection every 3 weeks for a minimum of 4 doses and a maximum of 12 doses. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion every 3 weeks, with a maximum of 12 doses. Vigil was administered first, followed 30 minutes later by atezolizumab. 1 cycle = 21 days
- Part 3: Atezo: Participants continue on single agent atezolizumab until disease progression. Atezolizumab was administered at a dose of 1200 mg as an intravenous infusion. 1 cycle = 21 days.
Arm/Group | Part 1: Vigil + Atezo | Part 2: Vigil | Part 2: Atezo | Part 2: Vigil and Atezo | Part 3: Atezo
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/11 | 3/10 | 9/21 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/11 | 4/10 | 1/21 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 9/11 | 10/10 | 15/21 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Vigil + Atezo (N=3) | Part 2: Vigil (N=11) | Part 2: Atezo (N=10) | Part 2: Vigil and Atezo (N=21) | Part 3: Atezo (N=1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Partial Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weakness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased Creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Vigil + Atezo (N=3) | Part 2: Vigil (N=11) | Part 2: Atezo (N=10) | Part 2: Vigil and Atezo (N=21) | Part 3: Atezo (N=1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (6) | 2 (5) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goiter nodular (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 7 (8) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (5) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (8) | 2 (2) | 4 (6) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swallowing difficult (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema extremities (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 3 (6) | 7 (7) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Heat intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ALT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
BUN increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ST segment elevated (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Intermittent headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Anxiety reaction (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2) | 4 (4) | 3 (5) | 0 (0)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT03073525/Prot_SAP_001.pdf